CLINICAL TRIAL: NCT05491564
Title: SoftStitch™ for All-Inside Meniscal Repair: Comparative Analysis of Patient Reported Outcome Measures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AIRR-0065
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Meniscus Tear

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: SoftStitch™ — The SoftStitch™ meniscal repair system includes a unique knotless all-inside meniscal repair implant with all suture fixation, eliminating the traditional hard plastic PEEK anchors used in the previous devices.

SUMMARY:
Acute and traumatic knee meniscus tears are a frequent occurrence. Evidence shows meniscal repair results in more favorable patient reported outcomes and articular cartilage preservation.1 This prospective, multicenter, single cohort, longitudinal study is intended to evaluate the effectiveness and safety profile of SoftStitch™ when used as standard of care for All-Inside Meniscal Repair. Electronic Patient Reported Outcome Measures (ePROM), functional assessments of the knee, Adverse Events of interest and Adverse Device Effects will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed meniscal tear by physical exam and MRI (minimum 1.5T)
2. Recommended to undergo surgical intervention using SoftStitch™ for All-Inside meniscus repair of longitudinal tears on the posterior horn that a surgeon would traditionally repair with two or more all-inside devices, as standard of care
3. Normal mechanical alignment; < 5° varus and < 7° valgus, of the affected knee by clinical assessment or X-Rays
4. Male or female, ≥ 18 years old and ≤55
5. Provide written informed consent
6. Able and willing to participate in follow up visits
7. Have a valid email and internet access to receive and respond to ePROs throughout the study

Exclusion Criteria:

1. Meniscal tears which are not amendable to repair, such as degenerative, flap, radial, complex, etc.
2. ACL-injured knees that are unstable (concomitant ACL reconstruction OK to include)
3. Sensitivity to silicone, polyester, nylon, FD&C Blue No. 2 dye and beeswax
4. Blood supply limitations and previous or active6, joint or systemic, infections which may decrease healing
5. Skeletally immature defined as patients with open epiphyseal plates viewed on radiographs
6. Concomitant disease that would interfere with study outcomes
7. Congenital ligamentous hypermobility defined by Beighton score 4 or 5
8. Locked knee or haemarthrosis7
9. Mutiligament injuries requiring multiligament surgical stabilization
10. Concomitant hybrid meniscal repair techniques or devices
11. Advanced Osteoarthritis; Kellgren Lawrence ≥ 2
12. Fracture of the lower extremities within 6 months prior to screening
13. Previous surgery on the affected knee within 12 months prior to screening
14. Subject is included in a vulnerable population (child, prisoner, etc).
15. Subject is requesting or receiving Worker's compensation related to the knee injury
16. Inability to reply to online questionnaires because of mental impairment
17. Participation in another clinical investigation in the next two years

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Individuals recommended to undergo meniscal repair using SoftStitch™ in routine clinical practice will be considered for participation in this study.
  50 subjects, male and female, ≥ 18 years old who have been legally consented and meet the eligibility criteria will be enrolled at the time of surgery.
  Subjects will be recruited from the principal investigator's patient population or referrals from other physicians.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Lysholm Score | Collected at baseline, 6 weeks, 3 months post-op, 6 months post-op, 12 months post-op, and 24 months post-op. The changes from baseline will be assessed.
  It is a condition specific scoring system to provide the patient perspective of their illness. The Lysholm scoring scale currently consist of eight domains that measure: pain, instability, locking, swelling, limp, stair climbing, squatting, and need for support. The total score is the sum of all responses and ranges from 0-100 points with 95 to 100 as excellent outcome, 84 to 94 as good outcome, 65 to 83 as fair outocome and <65 as poor outcome.
Tegner Activity Scale | Collected at baseline, 6 weeks post-op, 3 months post-op, 6 months post-op, 12 months post-op, and 24 months post-op. The changes from baseline will be assessed.
  It is a numerical scale that ranges from 0 - 10 to measure the ability to perform specific activities. An activity level of 5 to 10 is recorded only if the patient participates in competitive or recreational sports. That is, an activity level of 10 corresponds to participation in competitive sports such as soccer, football, and rugby at the elite level; an activity level of 6 points corresponds to participation is recreational sports. An activity level of 0 is assigned if a person is on sick leave or receiving a disability pension because of knee problems.
International Knee Documentation Committee (IKDC) Subjective Measure | Collected at baseline, 6 weeks post-op, 3 months post-op, 6 months post-op, 12 months post-op, and 24 months post-op. The changes from baseline will be assessed.
  The IKDC is a knee-specific subjective scale rather than a disease-specific measure. The IKDC to measure change in symptoms, sports activity, and function in patients with diverse knee conditions. The symptoms subscale evaluates pain, stiffness, swelling and giving-way of the knee. The sport activity subscale measures functions such as going up and down the stairs, rising from a chair, squatting and jumping. The knee function subscale asks the subject how well does the knee work now and before the injury. Individual scores are added and then transformed to a scale ranging from 0 to 100. The calculated IKDC score should be interpreted as a measure of function, such that high scores represent high levels of function and lower levels of symptoms. The instrument has demonstrated reliability and validity to measure patient reported outcomes.
Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 | Collected at baseline, 6 weeks post-op, 3 months post-op, 6 months post-op, 12 months post-op, and 24 months post-op. The changes from baseline will be assessed.
  It is a ten-item global health questionnaire developed by the National Institutes of Health (NIH) to assess health-related quality of life compared with normal values in the U.S. general population. It measures five domains: physical function, fatigue, pain, emotional distress, and social health on a five-point response matrix. Nine of ten questions are answered using 5-point Likert scales, and the 10th question is answered using a numerical rating scale. The questionnaire does not yield an overall score but gives physical and mental health component scores that are transformed to t-score distributions with a mean of 50 and standard deviation of 10. The structure of the score should offer greater responsiveness to changes in general health. Responsiveness is defined as the ability of an instrument to measure change over time.
McMurray Test | Collected at baseline, 6 months post-op, 12 months post-op, and 24 months post-op. The changes from baseline will be assessed.
  It was designed to detect tears in the posterior segment of the meniscus. It is performed by placing the knee beyond 90° of flexion and then rotating the tibia on the femur into full internal rotation to test the lateral meniscus, or full external rotation to test the medical meniscus. The same movements are performed in gradually increasing degrees of knee flexion to progressively load more posterior segments of the menisci. No valgus or varus stress is applied. The surgeon will palpate the joint line medially and laterally. A positive test includes a thud or click that can sometimes be heard but can always be felt.